CLINICAL TRIAL: NCT06603610
Title: Adaptation and Implementation of an Intensive Geriatric Service Worker (IGSW) Model of Care for Socially Isolated Older Adults: a Pilot Randomized Trial
Brief Title: Adaptation and Implementation of an Intensive Geriatric Service Worker (IGSW) Model of Care for Socially Isolated Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-277
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Older Adults; Social Isolation
Keywords: older adults; social isolation
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Participants in this arm will receive the intervention.
  Interventions: Other: Intensive geriatric service worker model of care
- Control (Placebo Comparator): Participants in the control group will receive their usual care, along with a booklet containing information about locally available resources, such as those related to meal preparation, grocery delivery, housekeeping, pharmacies that deliver medicines, home care, and Wheel-Trans. Participants in this arm will also receive telephone follow-up support.
  Interventions: Other: Information brochure and telephone follow-up support

INTERVENTIONS:
Other: Intensive geriatric service worker model of care — Participants in the intervention group will receive care from an intensive geriatric service worker (IGSW), who will help the participant:
  (i) Coordinate community resources and actively support participants' instrumental activities of daily living (IADLs) (e.g., linking participants with Meals-on-Wheels, taking participants to appointments) (ii) Advocate for support from home care for completing activities of daily living (ADLs) (iii) Implement patients' prioritized treatment recommendations made by healthcare professionals (e.g., supporting patients to purchase and install home safety equipment because this aligns with their values and preferences).
  Arms: Intervention
Other: Information brochure and telephone follow-up support — Participants will be e-mailed or mailed a booklet containing information about locally available resources including (1) meal preparation, (2) grocery delivery, (3) housekeeping, (4) pharmacies that deliver medications, (5) home care, and (6) Wheel-Trans. Participants will receive a scripted phone call from the study research coordinator one and three months after study enrolment to see if they have questions about the booklet material.
  Arms: Control

SUMMARY:
In this study, participants will be randomly assigned to receive either the intervention or control treatment for up to 6 months. Participants in the intervention group will receive care from an intensive geriatric service worker (IGSW), who will help the participant:

(i) Coordinate community resources and actively support participants' instrumental activities of daily living (IADLs) (e.g., linking participants with Meals-on-Wheels, taking participants to appointments) (ii) Advocate for support from home care for completing activities of daily living (ADLs) (iii) Implement patients' prioritized treatment recommendations made by healthcare professionals (e.g., supporting patients to purchase and install home safety equipment because this aligns with their values and preferences).

Participants in the control group will receive their usual care, along with a booklet containing information about locally available resources, such as those related to meal preparation, grocery delivery, housekeeping, pharmacies that deliver medicines, home care, and Wheel-Trans.

We are interested in learning about the number and demographic characteristics of participants we will be able to recruit to the study, who will remain in the study and who will be adherent to their prioritized treatment recommendations. We are also interested in learning about changes in participants' quality of life, proportion of IADLs being completed independently or with support, emergency department visit rate, and hospitalization rate at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

(i) adults aged ≥65 years old (ii) socially isolated, defined as living alone (iii) identified by the multidisciplinary Acute Care of the Elderly team, Internal Consultation Team, or Elders' Clinic as having one or more instrumental activity of daily living (IADL) impairments (defined as per the Lawton IADL scale) that could be supported by the intensive geriatric service worker (iv) capable of consenting to study participation or have a substitute decision-maker who can provide consent on their behalf (v) able to understand and communicate in English (e.g., if a participant is hearing impaired, but they can lip read or hear sufficiently with a hearing aid, they will be included) or know someone who can help with translation (vi) living in a private dwelling (e.g., apartment, house, condominium) within a geographical catchment area (i.e., boundaries will be Bloor St, Don Valley Parkway, Lakeshore Blvd, and Yonge St) (vii) a patient of a family physician or nurse practitioner (or be willing to become a patient of a family physician or nurse practitioner).

Exclusion Criteria:

(i) live in a retirement home, long-term care home or shelter (because there is varying availability of resources to support patients' activities of daily living (ADLs) and IADLs in these settings and we want to implement the IGSW care model where we hypothesize that it will have the greatest impact (ii) do not have a fixed address (iii) are participating in another study (iv) are being transferred to a rehabilitation facility other than Providence Healthcare prior to discharge home (Providence Healthcare is a collaborating study site; our team has an ongoing research collaboration with the medical rehabilitation unit at Providence Healthcare [where ACE and ICT medical consultation patients are transferred]

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Implementation Feasibility | Between 3 months to 1 year
  The number of participants (i) recruited (over the entire 12-month recruitment period and per month), (ii) retained (remain in the IGSW care model until prioritized recommendations are implemented, are discharged from the program because they are admitted to a retirement or LTC home, or complete the intervention; number of participants in the control group who provide follow-up data at 3 and 6 months) (iii) fully adherent to patients' prioritized recommendations during the trial period (% full adherence to [a] all prioritized recommendations, [b] >75% of prioritized recommendations, and [c] ≥1 prioritized recommendation at 3 and 6 months) and (iv) sustained linkages to community agencies to provide ADL and IADL support (number of participants with linkages to [a] all community agencies, [b] ≥1 community agency at 3 and 6 months).

SECONDARY OUTCOMES:
Quality of Life | 3 and 6 months
  Change in quality of life will be measured with the EQ-5D-5L
Proportion of IADLs being completed independently or with support | 3 and 6 months
Emergency department visit rate | 3 and 6 months
Hospitalization rate | 3 and 6 months
Long-term care home admission rate | 3 and 6 months
Length of hospitalization | 6 months
  This will be measured for study participants admitted to hospital.

IPD SHARING:
Plan to Share IPD: No